CLINICAL TRIAL: NCT01421160
Title: A Pilot Study to Assess the Effects of Regulating Urine pH Levels for Alleviating Chronic Joint Pain
Brief Title: Regulating Urine pH Levels to Alleviate Chronic Joint Pain
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: PI left the institution prior to any data being collected
Sponsor: Texas Tech University Health Sciences Center, El Paso (Other)
Responsible Party: Principal Investigator, Dennis Miller, Assistant Professor, Texas Tech University Health Sciences Center, El Paso
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: citrate1
Record Dates: First submitted 2011-07-20; First posted 2011-08-22 (Estimated); Last update posted 2017-05-16 (Actual); Status verified 2017-05

CONDITIONS: Arthritis
Keywords: Chronic; Inflammatory; Joint; Pain
MeSH Terms: conditions — Arthritis; Bronchiolitis Obliterans Syndrome; Pain | interventions — Sodium Citrate; Citric Acid; Citrates

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: sodium citrate and citric acid — sodium citrate and citric acid equivalent to 1 mEq/ml bicarbonate (usual dose 10-30 mls/day diluted with water)
  Other Names: Cytra-2

SUMMARY:
This study aims to determine the causal relationship between regulating urine pH levels between 7.0 and 7.5 and decreasing chronic joint pain. The investigators hypothesize that maintenance of an alkaline urinary pH will result in a decrease in personally reported levels of chronic joint pain using a citrate treatment regimen.

DETAILED DESCRIPTION:
STUDY SYNOPSIS / Literature Review Inflammation is a local immune response to injury, infection and foreign molecules. Notwithstanding the provoking cause, inflammation is thought to have evolved as an adaptive response for restoring tissue homeostasis. The local inflammatory response causes acidosis and pain has been associated with induced acidosis of various origins - diet, injury, exercise, stress, medications, disease state or aging.

Inflammatory and degenerative joint diseases are major causes of chronic pain. In general, inflammatory causes (e.g. rheumatoid arthritis, RA) are more common in younger individuals, while degenerative causes (e.g. osteoarthritis, OA) are more often seen in the elderly [Schaible et al, 2009]. Pain perception is extremely complex and a perceived connection has been noted between the level of pain felt by individuals and bodily fluid hydrogen ion concentration, i.e. pH; oral water-soluble alkaline components containing K, Ca, Mg and Cl salts have been used for reducing bodily fluid and tissue acid concentrations. Urine pH is now considered to reflect the bodily acid-base balance and is directly related to the dietary acid-base load [Welch et al, 2008].

Currently, potassium citrate (Kcit, 45-60 mEq daily) has been widely used in urology for treatment of patients with uric acid and cystine stones [Sterrett et al, 2008; Spivacow et al, 2010]. Aside from the use of Kcit in the treatment of kidney stones, there have been isolated reports about the anti-inflammatory and hypoalgesic systems effects of Kcit. Alkalinization by diet alone has also been effective for removing uric acid from the body, though its effects on urine pH levels are weaker [Kanbara, Hakoda & Seyama, 2010]. It is considered that alkalinization of urine reflects body fluid alkalinization. This has the perceived effects of increased bone density, improved muscle function, and a speculative decrease in insulin resistance [Pizzorno, Frassetto & Katzinger, 2010].

Research Project Question/Theme The investigators aim to determine causal relationship between regulating urine pH levels between 7.0 and 7.5 and decreasing chronic joint pain. The investigators hypothesize that maintenance of an alkaline urinary pH will result in a decrease in personally reported levels of chronic joint pain using a citrate treatment regimen.

Project Design:

Subjects will be recruited from local physician's practices, primarily at TTUHSC clinics, by the Principal Investigator and the Co-Investigators. Subjects who report a presence of joint pain for more than six months, and meet the inclusion/exclusion criteria, will be eligible for participation.

Any Adverse Events (AEs) will be monitored by the Principal Investigator and Co-Investigators, and reported by the Study Coordinator to the IRB.

Subjects for the study will be identified by the Principal Investigator and Co-Investigators from local TTUHSC clinics.

After the subject agrees to participate and informed consent has been given, the study coordinator will explain the study procedures and baseline measurements will be assessed using diagnostic imaging and lab testing. All subjects will be asked to obtain and/or provide a copy of recent X-rays or an MRI of the affected joint and lab tests (CBC, liver and kidney panels). Images and tests must be recent and taken within the past 6 months of enrollment in the study.

After the baseline measurements have been established, instructions on the urine alkalinization treatment regimen will be distributed to the subject and treatment solution will be obtained. This treatment will vary from person to person and is easily modified.

Subjects will measure, report, and take the treatment for 6 months.

While on the treatment, all subjects will be asked to report and/or measure the following values on a daily basis:

* Report when and how much treatment was taken that day
* Measure urine pH levels daily at 10 A.M. using a pH strip
* Rate their pain 3X daily using a modified pain rating scale
* Report daily food and beverage intake
* Visit the physician investigator for monthly a follow-up visit to review the pain ratings and pH values noted during the past month

Analysis:

Using the SAS System, the investigators calculated the minimum number of enrolled subjects that is required to achieve statistical results is 21. The investigators estimated that a minimum number of 16 subjects must complete the study in order to achieve sufficient, statistically powerful results. In order to ensure successful completion of the statistical data analysis, the investigators decided to enroll twice the minimum number of subjects required (16x2) and will enroll a total of 32 subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Presence of joint pain of perceived inflammatory and non-inflammatory origin for more than six months. More specifically:

   * Subjects with osteoarthritis (OA) of the knee will be preferred for inclusion in this study.
   * Subjects with other joint pain history will be included pursuant on approval from Dr. Miller or Dr. Pema.
2. Age 21 to 80 years old and otherwise in good health (excluding the joint pain).
3. Able to understand and comply with the assigned urine alkalinization instructions.
4. Has a working and reliable telephone number for continued contact as necessary during the study.
5. Ability to obtain X-rays of the affected joint. Imaging of the painful joint will be necessary at the beginning of the study for baseline considerations; if images from the last 6 months are available, no new imaging would be necessary.
6. Ability to obtain lab tests (Complete Blood Count and Comprehensive Metabolic Panel) or can obtain documentation of recent lab tests that have been taken within one month prior to enrollment.
7. Ability to obtain lab tests at 3 and 6 months during participation in the study.

Exclusion Criteria:

1. Presence of joint pain with known joint osseous changes.
2. Pregnant or lactating women will not be enrolled in the study.
3. Positive medical history of:

   * Diabetes
   * Neuropathies
   * Gout
   * Psychiatric diseases and conditions, including anxiety, depression, PTSD, distress
   * Psychosocial abnormalities
   * Dementia or other memory disturbances
   * Alcoholism or substance abuse
   * Renal failure and/or abnormal renal function (kidney disease or dysfunction). Specifically, Creatinine (Creat) values that are over 1.2mg/dL and Urea Nitrogen (BUN) values that are over 22mg/dL are considered abnormal.
   * No history of cardiovascular disease, intestinal angina or arrhythmias
   * No history of sodium restrictions
   * Pt. should not be taking medications which produce pain such as angiotensin converting enzyme (ACE) inhibitors and Statins (Lisinopril, Quinapril, Ramipril)
4. Does not have reliable telephone communication.
5. Does not have the ability to obtain an X-ray and does not have the ability to obtain documentation of a recent X-ray within the last six months.
6. Does not have the ability to obtain lab tests (Complete Blood Count and Comprehensive Metabolic Panel) and does not have the ability to obtain documentation of recent lab tests that have been taken within one month prior to enrollment.
7. Does not have the ability to obtain lab tests at 3 and 6 months during participation in the study.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-07; Primary Completion 2012-03 (Estimated); Study Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
Pre-and post test pain rating | Six months
  At the beginning of the study, during office visits, and at the end of the study, subjects will be asked to visually and numerically rate their pain levels.
Change in Urine pH from baseline | Six months
  Subject's daily self-report of this measure will be provided to study investigator at each office visit.
Changes in lab results (routine blood work) from baseline | Six months.
  Assessed at the beginning, middle (3 months) and end of the six month study.
Change in amount of alkalization medication taken daily | Six months
  Subject's daily self-report of this measure will be provided to study investigator at each office visit.

SECONDARY OUTCOMES:
Daily food and beverage intake | Six months
  Subject's daily self-report of this measure will be provided to the study investigator at each office visit.

CONTACTS AND LOCATIONS:
Overall Officials: Dennis W Miller, MD, Principal Investigator — Department of Anesthesiology; Texas Tech University Health Sciences Center; Paul L. Foster School of Medicine
Locations (1):
- Department of Anesthesiology; Texas Tech University Health Sciences Center; Paul L. Foster School of Medicine, El Paso, Texas, United States

REFERENCES:
- [Background] Schaible HG, Richter F, Ebersberger A, Boettger MK, Vanegas H, Natura G, Vazquez E, Segond von Banchet G. Joint pain. Exp Brain Res. 2009 Jun;196(1):153-62. doi: 10.1007/s00221-009-1782-9. Epub 2009 Apr 11. PMID 19363606
- [Background] Goldring MB, Goldring SR. Osteoarthritis. J Cell Physiol. 2007 Dec;213(3):626-34. doi: 10.1002/jcp.21258. PMID 17786965
- [Background] Devchand PR, Keller H, Peters JM, Vazquez M, Gonzalez FJ, Wahli W. The PPARalpha-leukotriene B4 pathway to inflammation control. Nature. 1996 Nov 7;384(6604):39-43. doi: 10.1038/384039a0. PMID 8900274
- [Background] Gurol et al, US Patent 2007/0218126 A1. Compositions and methods for reducing inflammation and pain associated with acidosis (7p.).
- [Background] Sterrett SP, Penniston KL, Wolf JS Jr, Nakada SY. Acetazolamide is an effective adjunct for urinary alkalization in patients with uric acid and cystine stone formation recalcitrant to potassium citrate. Urology. 2008 Aug;72(2):278-81. doi: 10.1016/j.urology.2008.04.003. Epub 2008 Jun 4. PMID 18533229
- [Background] Pizzorno J, Frassetto LA, Katzinger J. Diet-induced acidosis: is it real and clinically relevant? Br J Nutr. 2010 Apr;103(8):1185-94. doi: 10.1017/S0007114509993047. Epub 2009 Dec 15. PMID 20003625
- [Background] Kiwull-Schone H, Kiwull P, Manz F, Kalhoff H. Food composition and acid-base balance: alimentary alkali depletion and acid load in herbivores. J Nutr. 2008 Feb;138(2):431S-434S. doi: 10.1093/jn/138.2.431S. PMID 18203917
- [Background] Kanbara A, Hakoda M, Seyama I. Urine alkalization facilitates uric acid excretion. Nutr J. 2010 Oct 19;9:45. doi: 10.1186/1475-2891-9-45. PMID 20955624
- [Background] Welch AA, Mulligan A, Bingham SA, Khaw KT. Urine pH is an indicator of dietary acid-base load, fruit and vegetables and meat intakes: results from the European Prospective Investigation into Cancer and Nutrition (EPIC)-Norfolk population study. Br J Nutr. 2008 Jun;99(6):1335-43. doi: 10.1017/S0007114507862350. Epub 2007 Nov 28. PMID 18042305
- [Background] Medzhitov R. Origin and physiological roles of inflammation. Nature. 2008 Jul 24;454(7203):428-35. doi: 10.1038/nature07201. PMID 18650913
- [Background] Basbaum AI, Bautista DM, Scherrer G, Julius D. Cellular and molecular mechanisms of pain. Cell. 2009 Oct 16;139(2):267-84. doi: 10.1016/j.cell.2009.09.028. PMID 19837031
- [Background] Aras B, Kalfazade N, Tugcu V, Kemahli E, Ozbay B, Polat H, Tasci AI. Can lemon juice be an alternative to potassium citrate in the treatment of urinary calcium stones in patients with hypocitraturia? A prospective randomized study. Urol Res. 2008 Dec;36(6):313-7. doi: 10.1007/s00240-008-0152-6. Epub 2008 Oct 23. PMID 18946667
- [Background] McNally MA, Pyzik PL, Rubenstein JE, Hamdy RF, Kossoff EH. Empiric use of potassium citrate reduces kidney-stone incidence with the ketogenic diet. Pediatrics. 2009 Aug;124(2):e300-4. doi: 10.1542/peds.2009-0217. Epub 2009 Jul 13. PMID 19596731
- [Background] Whitson PA, Pietrzyk RA, Jones JA, Nelman-Gonzalez M, Hudson EK, Sams CF. Effect of potassium citrate therapy on the risk of renal stone formation during spaceflight. J Urol. 2009 Nov;182(5):2490-6. doi: 10.1016/j.juro.2009.07.010. Epub 2009 Sep 17. PMID 19765769
- [Background] Spivacow FR, Negri AL, Polonsky A, Del Valle EE. Long-term treatment of renal lithiasis with potassium citrate. Urology. 2010 Dec;76(6):1346-9. doi: 10.1016/j.urology.2010.02.029. PMID 20399488
- [Background] Iakovenko EP, Agafonova NA, Pokhal'skaia OIu, Kolganova AV, Nazarbekova RS, Ivanov AN, Davletshina IV, Popova EV, Prianishnikova AS, Ovchinnikova NI, Iakovenko AV, Aldiiarova MA, D'iachkoava AV, Gioeva IZ. [The use of bismuth tripotassium dicitrate (De-Nol), a promising line of pathogenetic therapy for irritated bowel syndrome with diarrhea]. Klin Med (Mosk). 2008;86(10):47-52. Russian. PMID 19069460
- [Background] Balkowiec-Iskra E. [The role of immune system in inflammatory pain pathophysiology]. Pol Merkur Lekarski. 2010 Dec;29(174):395-9. Polish. PMID 21298993